CLINICAL TRIAL: NCT03102775
Title: A Cluster-randomised Study Evaluating the Effectiveness of a Skill-training Programme for Social Work Professionals for Improving the Follow-up of Low Income Families Within Norwegian Welfare Services
Brief Title: Comprehensive Follow-up of Low Income Families. A Cluster-randomized Study
Acronym: CRCT-HOLF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo Metropolitan University (Other)
Collaborators: Norwegian Labour and Welfare Administration (Other)
Responsible Party: Principal Investigator, Ira Malmberg-Heimonen, Professor, Soc Sci dr., Oslo Metropolitan University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 48510 (nsd)
Record Dates: First submitted 2017-03-07; First posted 2017-04-06 (Actual); Last update posted 2022-09-27 (Actual); Status verified 2022-09

CONDITIONS: Poverty
Keywords: poverty; unemployment; cluster-randomized; family-project

STUDY DESIGN:
Intervention Model Description: Cluster-randomized study. After baseline at office leader and family coordinator level as well as administrative data for families in target group, offices have been randomized to experimental and control group offices. The HOLF-model is implemeted in experimental group offices, while control group offices implement local family projects. Effects on families are analysed on the four main follow-up areas: employment, housing, financial situation and the social situation of the children.
Who Masked: Participant
Masking Description: While the leaders and family-coordinators are aware of whether the office has been randomized to experimental or control group offices, the families are masked for this information. they are only aware of participating in a family project, but not if experimental or control condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Comprehensive follow-up program (Experimental): 15 offices have been randomized to experimental group. Experimental group offices implement the HOLF model developed by the Labor and Welfare Administration
  Interventions: Other: Comprehensive follow-up program for low-income families
- Local family projects (Active Comparator): 14 offices have been randomized to control group. these implement local family projects. These are developed based on local practice needs
  Interventions: Other: local family projects

INTERVENTIONS:
Other: Comprehensive follow-up program for low-income families — The main follow-up areas within the HOLF-program is to improve employment, housing, financial situation of the children. Beside manuals, family coordinators participate in five seminars with home-based tasks in between. Alo a comprehensive supervision structure is implemented that follow the train the trainer model. Coordinators ought to work directly with th families, but also with other actors important to the family, such as child-welfare and school. Coordinators should use specific tools improving the quality of the meetings, such as forms for preparation of meetings, being goal-focused and empowering.
  Arms: Comprehensive follow-up program
Other: local family projects — The control group offices will develop local family projects, depending on local needs. they will also recruit and follow-up families.
  Arms: Local family projects

SUMMARY:
In a cluster-randomized design, the study evaluates the effectiveness of a skill- training program for social work professionals with the aim of improving the follow-up of low income families within Norwegian labor and welfare services. While the Norwegian Labor and Welfare Administration are responsible for developing and implementing the program, researchers at Oslo and Akershus University College are conducting an independent evaluation of its effectiveness. By close follow up and better coordination of existing services the model aims to improve the financial and housing situation of the family, labor market attachment among the parents and the social inclusion of children. The cluster-randomized field experiment will take place over a 40-month period, involving 29 labor and welfare offices, 58 family coordinators and, based on estimations, 650 families. The research is funded by the Norwegian Labor and Welfare Administration.

The project is financed by Labour and Welfare Administration and led by Ira Malmberg-Heimonen, Faculty of Social Sciences. Participants in the project are: Ira Malmberg-Heimonen (project leader), Anne Grete Tøge, Krisztina Gyüre, Knut Fossestøl, Marianne Rugkåsa, Berit Bergheim and Tone Liodden.

DETAILED DESCRIPTION:
Comprehensive follow up of low-income families. A cluster-randomised study. Start 1.1 2016, Finnish 31.5 2019 Funding: Norwegian Labour and Welfare Administration

Collaboration:

Norwegian Labour and Welfare Administration

Labour and Welfare offices:

NAV Alna, NAV Asker, NAV Bergenhus, NAV Bjerke, NAV Bodø, NAV Bærum, NAV Elverum, NAV Fana, NAV Frogner, NAV Gamle Oslo, NAV Gjøvik, NAV Grunerløkka, NAV Halden, NAV Harstad, NAV Haugesund, NAV Horten, NAV Larvik, NAV Lerkendal, NAV Lillehammer, NAV Malda, NAV Moss, NAV Nordstrand, NAV Rana, NAV Ringsaker, NAV Sandefjord, NAV Sandnes, NAV Skedsmo, NAV St.Hanshaugen, NAV Værnes

International collaborators:

Professor Jukka Vuori, Finnish Institute of Occupational Health, Finland Professor Richard Price, University of Michigan, US Senior researcher Gayle Hamilton, MDRC New York, US Professor Bruce Thyer, Florida State University, US

The Norwegian Labour and Welfare Administration has developed a comprehensive model in order to improve the follow-up of low income families, and thereby decrease poverty and its consequences. By close follow up and better coordination of existing services the model aims to improve the financial and housing situation of the family, labour market attachment among the parents and the social inclusion of children.

Oslo and Akershus University College has been commissioned to evaluate the effects of the model between 2016 to 2019, with long-term follow-ups until 2021. The evaluation is conducted as a cluster-randomized controlled trial, where 29 labor and welfare offices have been randomly assigned to the experimental and control group. All 29 offices receive funding two family coordinators each in order to work with low-income families. While the experimental group offices implement the HOLF-model for the follow-up of low income families, the control group offices implement locally developed models.

Prior to randomization, a baseline questionnaire was collected from office leaders and family-coordinators, while baseline information on families is collected based on administrative data prior to randomization and questionnaire data after randomization, but prior taking part in family projects. Shorter-term effects will be measured + 12 months after baseline for families, and long-term effects will be measured based on administrative data fup to four years after baseline.

Researchers at Oslo and Akershus University College analyses the implementation processes and effects of the implementation through questionnaires, administrative data, observational data, qualitative interviews with leaders, family coordinators and families.

The project will contribute to increased knowledge about measures to improve the follow up of low income families. It will generate knowledge of whether the HOLF-model is more effective than locally developed follow-up models, knowledge important for the discussion of evidence-informed vs practice-based interventions.

The project is financed by Labor and Welfare Administration and led by Ira Malmberg-Heimonen, Faculty of Social Sciences.

Participants in the project are: Ira Malmberg-Heimonen (project leader), Anne Grete Tøge, Krisztina Gyüre, Knut Fossestøl, Marianne Rugkåsa, Berit Bergheim and Tone Liodden.

ELIGIBILITY:
Inclusion Criteria:

Each of the 29 offices identified a target group of families prior to randomization based on the following characteristics:

* reliance on social assistance as a main source of income at least for six of the latest 12 months, or
* received social assistance in addition to other types of welfare support at least for six of the latest 12 months, and
* have up to four children under the age of 16. Based on these criteria offices identified a total of 3201 families.

Exclusion Criteria:

Families were excluded from participation in the project if:

* they participate in other comprehensive family projects
* one or both parents/caregivers are under treatment because of heavy substance abuse and/or serious mental disorders
* the child or the children are temporary placed in child welfare institutions or living with relatives or other caregivers.
* the family is under investigation by child welfare authorities, due to suspected child neglect or that a placement to new caregivers is in process.

Based on these criteria 320 families were excluded.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 884 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Changes in the employment situation from baseline to follow-ups | T2 (+12 months after baseline), T3 (+24 months) T4 (+36 months) -T5 (+48 months)
  Percentage employed
Change in the housing situation between baseline and follow-up | T2 (+12 months after baseline)
  Objective and subjective estimations of housing quality
Change in the financial situation between baseline and follow-ups | T2 (+12 months after baseline), T3 (+24 months) T4 (+36 months) T5 (+48 months)
  Income per month at follow-ups
Change in children's situation from baseline to follow-up | T2 (+12 months)
  Participation in kindergarden and other free-time activities

SECONDARY OUTCOMES:
Change in professional competence between baseline and follow-up | T2 (+18 months)
  Family coordinators professional competence. A six-item scale
Change in the level of working alliance between baseline and follow-up | T2 (+18 months)
  Working Alliance Inventory Scale (short version)

OTHER OUTCOMES:
Changes in leaders competence between baseline and follow-up | T2 (+18 months)
  Scale measuring office leaders competence in the follow-up of low-income families.

CONTACTS AND LOCATIONS:
Locations (29):
- Norway (29):
  - NAV Asker, Asker
  - NAV Bærum, Baerum
  - NAV Bergenhus, Bergen
  - NAV Fana, Bergen
  - NAV Bodø, Bodø
  - NAV Elverum, Elverum
  - NAV Gjøvik, Gjøvik
  - NAV Halden, Halden
  - NAV Harstad, Harstad
  - NAV Haugesund, Haugesund
  - NAV Horten, Horten
  - NAV Larvik, Larvik
  - NAV Lillehammer, Lillehammer
  - NAV Skjedsmo, Lillestrøm
  - NAV Rana, Mo i Rana
  - NAV Moss, Moss
  - NAV Alna, Oslo
  - NAV Bjerke, Oslo
  - NAV Frogner, Oslo
  - NAV Gamle Oslo, Oslo
  - NAV Gruneløkka, Oslo
  - NAV Nordstrand, Oslo
  - NAV St. Hanshaugen, Oslo
  - NAV Ringsaker, Ringsaker
  - NAV Sandefjord, Sandefjord
  - NAV Sandnes, Sandnes
  - NAV Madla, Stavanger
  - NAV Lerkendal, Trondheim
  - NAV Værnes, Værnes

IPD SHARING:
Plan to Share IPD: No
After embargo + 5 years after finishing study (2026)

REFERENCES:
- See also: homepage for the study — https://www.oslomet.no/forskning/forskningsprosjekter/holf-prosjektet
- Available data/document: final report (Norwegian) — https://skriftserien.hioa.no/index.php/skriftserien/article/view/649